CLINICAL TRIAL: NCT01517854
Title: Revatio Portal-Pulmonary Arterial Hypertension Trial (RePo1 Trial): A Randomized, Double-blinded, Placebo-controlled, Multi-center Study to Evaluate the Effects of Sildenafil Citrate (Revatio) 20 mg TID on Patients With Portal Pulmonary Arterial Hypertension (PPAH)
Brief Title: Revatio Portal-Pulmonary Arterial Hypertension Trial
Acronym: RePo1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RePo1
Record Dates: First submitted 2011-12-14; First posted 2012-01-25 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Portopulmonary Hypertension
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Revatio (Active Comparator)
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — 20 mg Revatio (sildenafil citrate) three times a day
  Arms: Revatio
Drug: Placebo — Placebo identical to Revatio (sildenafil citrate) three times a day
  Arms: Placebo

SUMMARY:
The investigators propose the first prospective, double blind, randomized controlled trial of treatment for pulmonary arterial hypertension (PAH) related to underlying portal hypertension. Specifically the investigators will evaluate the potential efficacy and safety of sildenafil (Revatio) in a 16 week blinded, multicentre study.

DETAILED DESCRIPTION:
PAH is a recognized complication of portal hypertension - termed portal-pulmonary hypertension (PPHTN). In the World Health Organization (WHO) classification PPHTN is categorized as a WHO group 1 condition. This categorization is appropriate as PPHTN shares similar pathological features and clinical presentation and as idiopathic (primary) pulmonary arterial hypertension (PAH). Advances in oral therapies in PAH (idiopathic, connective tissue disease, congenital heart disease) has deferred the need for parenteral therapies, lung transplantation and led to improvements in functional capacity, quality of life and survival. However unlike other forms of PAH, treatment options have not been formally evaluated for PPHTN and there are no approved medical therapies. Patients are unable to pay for medications. Consequently patients continue to endure the natural progression of PAH - a state characterized by progressive right heart failure, disability and death. Furthermore the unacceptable mortality associated with liver transplantation in the presence of hemodynamically significant PAH, leaves them with no therapeutic options. Therefore, new treatment options need to be systematically evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with PPHTN.
* A 6MWD test between 150 m and 450 m.
* A pulmonary vascular resistance (PVR) >250 dyn*sec*cm-5, a mean pulmonary artery pressure (PAPmean) ≥25 mmHg due to portal hypertension, and PCWP ≤ 15 mmHg. Right-heart catheterization results for the definite diagnosis of PH must follow the 2 - 6 week pre-treatment phase and not be older than 6 weeks at study start (will be considered as baseline values).
* Portal hypertension defined either clinically or hemodynamically by the presence of cirrhosis (by ultrasound or biopsy) or portal vein thrombosis / obstruction (proven by portal vein Doppler) and any one of the following within one year of entry into the study: 1) Ascites (on ultrasound of the abdomen); 2) Splenomegaly (on ultrasound of the abdomen); 3) Esophageal or Gastric Varices (proven endoscopically); 4) Hepatic-venous pressure gradient (HVPG) > 12 mmHg.
* Treatment naive patients (with respect to PAH specific medication) and patients. Prior use of sildenafil for erectile dysfunction will be permitted.
* 18 to 75 years of age at Visit 1.
* Patients who are able to understand and follow instructions and who are able to participate in the study for the entire period.
* Patients must have given their written informed consent to participate in the study after having received adequate previous information and prior to any study-specific procedures.

Exclusion Criteria:

* Participation in another clinical trial during the preceding 3 months.
* Pregnant women or breast feeding women.
* Patients with a medical disorder, condition, or history of such that would impair the patient's ability to participate or complete this study in the opinion of the investigator or the sponsor.
* Patients with a history of severe allergies or multiple drug allergies.
* Patients with hypersensitivity to the investigational drug or inactive constituents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-11-14 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in PVR after 16 weeks of treatment | 16 weeks

SECONDARY OUTCOMES:
For patients with a PVR>450 dynes/sec/cm5 at baseline, number of patients who have PVR below 350 dynes/sec/cm5 after 16 weeks of study drug will be determined | 16 weeks
Hospitalizations | 16 weeks
Death | 16 weeks
Complications of liver disease | 16 weeks
MELD score | 16 weeks
Renal dysfunction | 16 weeks
Desaturation | 16 weeks
Change in 6MWD from baseline | 16 weeks
Change in baseline WHO functional class | 16 weeks
Change in Brain Natruretic Peptide (BNP) from baseline | 16 weeks
Change from baseline in CAMPHOR and SF-36 measures of quality of life | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John T Granton, Study Chair — University Health Network, Toronto
Locations (3):
- Canada (3):
  - Lawson Health Research Institute (London Health Sciences Centre Research Inc.), London, Ontario
  - University Health Network, Toronto, Ontario
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec